CLINICAL TRIAL: NCT03617497
Title: Prevalence of Epilepsy and Sleep Wake Disorders in Alzheimer Disease
Acronym: PESAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Dr W Van Paesschen, Professor Doctor, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: S61745
Record Dates: First submitted 2018-07-24; First posted 2018-08-06 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer Disease; Alzheimer Dementia; Epilepsy; Sleep Wake Disorders
Keywords: Alzheimer Disease; Alzheimer dementia; Epilepsy; Sleep Wake Disorders; EEG; Polysomnography; Foramen ovale electrodes
MeSH Terms: conditions — Alzheimer Disease; Epilepsy; Sleep Wake Disorders | interventions — Polysomnography

STUDY DESIGN:
Intervention Model Description: The investigators will perform 48-hour ambulatory scalp-EEG and polysomnography in 100 participants with Alzheimer disease and 30 age-and gender-matched healthy participants. The investigators will determine the prevalence of 1.) epileptic discharges and epileptic seizures, 2.) sleep wake disorders and 3.) the interaction of epilepsy and sleep wake disorders in these two groups. A subgroup of 15 of these 100 participants with Alzheimer disease, with interictal epileptic spikes or sleep wake disorders (e.g., frequent nocturnal awakenings) will be invited to undergo an invasive EEG study with foramen ovale electrodes to determine the prevalence of hippocampal seizures, which are usually clinically silent and not detected with scalp EEG.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control participants (Active Comparator): Age- and gender matched healthy participant (n=30) with no cognitive problems and normal amyloid PET scan will undergo 48 hour scalp EEG and polysomnography
  Interventions: Diagnostic Test: scalp EEG and polysomnography
- Alzheimer disease (Active Comparator): Participants with Alzheimer disease (n=100) will undergo 48 hour scalp EEG and polysomnography
  Interventions: Diagnostic Test: scalp EEG and polysomnography
- Alzheimer disease with high seizure risk (Experimental): Selected participants with Alzheimer disease, with higher risk for silent hippocampal seizures after 48 hour scalp EEG and polysomnography (e.g. presence of interictal spikes or frequent nocturnal awakenings) (n=15) will undergo scalp EEG with foramen ovale electrodes with polysomnography
  Interventions: Diagnostic Test: scalp EEG and polysomnography; Diagnostic Test: scalp EEG with foramen ovale electrodes with polysomnography

INTERVENTIONS:
Diagnostic Test: scalp EEG and polysomnography — 48 hour 22 channel EEG with polysomnography
Diagnostic Test: scalp EEG with foramen ovale electrodes with polysomnography — long-term scalp EEG with additional foramen ovale electrodes with polysomnography
  Arms: Alzheimer disease with high seizure risk

SUMMARY:
Alzheimer disease is the most common of the neurodegenerative diseases. Epilepsy and sleep wake disorders are co-morbid conditions of Alzheimer disease. The investigators propose a prospective study using long-term EEG monitoring in combination with polysomnography to determine prevalence of epilepsy and sleep wake disorders in Alzheimer disease, and correlate these findings with clinical data, Alzheimer disease biomarkers and imaging studies (MRI and amyloid/tau-PET). In selected patients, the investigators will perform EEG studies with foramen ovale electrodes. The ultimate goal is to improve the outcome of patients with Alzheimer disease by early treatment of epilepsy and restoring sleep-wake disturbances.

DETAILED DESCRIPTION:
Alzheimer disease is the most common of the neurodegenerative diseases. Epilepsy and sleep wake disorders are co-morbid conditions of Alzheimer disease, and there is evidence to suggest that the interactions are bidirectional. Neuronal activity promotes the production and secretion of amyloid β, which could actually drive pathogenesis early in the course of Alzheimer disease, and has been described in sleep wake disorders and epilepsy. Epileptic seizures in Alzheimer disease are often subtle, nocturnal and easily overlooked. We propose a prospective study using long-term EEG monitoring in combination with polysomnography to diagnose epilepsy and sleep wake disorders in Alzheimer disease, and correlate these findings with clinical data, Alzheimer disease biomarkers and imaging studies (MRI and amyloid/tau-PET). It is the hypothesis of the investigators that participants with Alzheimer disease and interictal spikes or specified sleep wake disorders (e.g., frequent nocturnal awakenings) during 48 hour scalp EEG and polysomnography are at risk for having hippocampal seizures, which are often clinically silent and not detected on scalp EEG. The investigators will invite 15 of these participants to undergo EEG studies with foramen ovale electrodes to determine the prevalence of these hippocampal seizures. The ultimate goal is to improve the outcome of patients with Alzheimer disease by early treatment of epilepsy and restoring sleep-wake disturbances.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand the nature of the study and has the opportunity to have any questions answered. The participant has voluntarily signed the independent Review Board (IRB)/independent Ethics Committee (IEC) approved Informed Consent, prior to the conduct of any study procedures. If the participant is not fully competent, full informed consent must be obtained from a representative and assent must be obtained from the participant.
2. Participant who meets the National Institute on Aging and the Alzheimer's Association (NIA-AA) clinical criteria for mild cognitive impairment or probable Alzheimer Disease, and have:

   * Clinical Dementia Rating (CDR)-Global Score of 0.5
   * A Mini-Mental State Examination (MMSE) score of 22 to 30
   * Repeatable Battery for the Assessment of Neuropsychological Status-Delayed Memory Index (RBANS-DMI) score of 85 or lower
3. Participant has a positive amyloid Positron Emission Tomography (PET) scan.
4. Participant has a Modified Hachinski Ischemic Scale (MHIS) score of ≤ 4.
5. Participant has an identified, reliable, study partner (e.g., family member), who has frequent contact with the participant and who will provide information as to the participant's cognitive and functional abilities.

Exclusion Criteria:

1. Participant has evidence of any other clinically significant neurological disorder other than Alzheimer disease, including but not limited to:

   * Parkinson's disease
   * vascular dementia
   * significant cerebrovascular abnormalities
   * frontal-temporal dementia
   * Huntington's disease
   * normal pressure hydrocephalus
   * brain tumor
   * progressive supranuclear palsy
   * seizure disorder
   * subdural hematoma
   * multiple sclerosis
   * history of significant head trauma followed by persistent neurologic deficits
   * known structural brain abnormalities
   * obstructive sleep apnea syndrome treated with continuous positive airway pressure (CPAP)
2. Participant has a screening MRI scan, interpreted by a radiologist with evidence of infection, infarction (including multiple lacunas in a critical memory structure), or other focal lesions.
3. Participant has a history of or currently has schizophrenia, schizoaffective disorder or bipolar disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM)-V or International Classification of Diseases (ICD)-10 criteria.
4. Participant has a current diagnosis or history of drug or alcohol abuse (by DSM-V criteria) within 24 months prior to the study.
5. Participant has a history or evidence of a malignancy within the 2 years prior to the study.
6. Participant has a known history of Human Immunodeficiency Virus (HIV) infection.
7. Participant has had surgery under general anesthesia within 3 months prior to the study.
8. Receipt of an investigational product within a time period equal to 5 half-lives, if known, or within 6 weeks (for small molecules) or 6 months (for monoclonal antibodies or other biologics) prior the study.
9. Participant has any history of prior receipt of active immunotherapy directed against tau or amyloid.
10. Participant is taking anti-epileptic drugs or benzodiazepines.
11. Participant has an abnormally low vitamin B 12 (cobalamin), abnormal thyroxine (T4) or an abnormally high thyroid stimulating hormone (TSH) that is considered clinically significant by the investigator.
12. Subject has any visual, auditory or other impairment that in the Investigator's opinion would preclude collection of outcome measures.
13. In the opinion of the investigator, the subject has any clinically significant or uncontrolled medical or psychiatric illness, or has had an infection requiring medical intervention in the past 30 days.
14. Subject has had a myocardial infarction, unstable angina, stroke, transient ischemic attack or required intervention for any of these conditions (e.g., coronary artery bypass graft, percutaneous coronary intervention via cardiac catheterization, thrombolytic therapy), within 6 months of the study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Epilepsy | during EEG recording
  presence of epileptic activity
Sleep wake disorder | during polysomnographic recording
  presence of sleep wake disorders

CONTACTS AND LOCATIONS:
Overall Officials: Wim Van Paesschen, MD PhD, Principal Investigator — UZ and KU Leuven
Locations (1):
- University Hospitals Leuven, department of Neurology, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Ju YE, Lucey BP, Holtzman DM. Sleep and Alzheimer disease pathology--a bidirectional relationship. Nat Rev Neurol. 2014 Feb;10(2):115-9. doi: 10.1038/nrneurol.2013.269. Epub 2013 Dec 24. PMID 24366271
- [Background] Musiek ES, Holtzman DM. Mechanisms linking circadian clocks, sleep, and neurodegeneration. Science. 2016 Nov 25;354(6315):1004-1008. doi: 10.1126/science.aah4968. PMID 27885006
- [Background] Ooms S, Overeem S, Besse K, Rikkert MO, Verbeek M, Claassen JA. Effect of 1 night of total sleep deprivation on cerebrospinal fluid beta-amyloid 42 in healthy middle-aged men: a randomized clinical trial. JAMA Neurol. 2014 Aug;71(8):971-7. doi: 10.1001/jamaneurol.2014.1173. PMID 24887018
- [Background] Noebels J. A perfect storm: Converging paths of epilepsy and Alzheimer's dementia intersect in the hippocampal formation. Epilepsia. 2011 Jan;52 Suppl 1(Suppl 1):39-46. doi: 10.1111/j.1528-1167.2010.02909.x. PMID 21214538
- [Background] Horvath A, Szucs A, Barcs G, Noebels JL, Kamondi A. Epileptic Seizures in Alzheimer Disease: A Review. Alzheimer Dis Assoc Disord. 2016 Apr-Jun;30(2):186-92. doi: 10.1097/WAD.0000000000000134. PMID 26756385
- [Background] Lam AD, Deck G, Goldman A, Eskandar EN, Noebels J, Cole AJ. Silent hippocampal seizures and spikes identified by foramen ovale electrodes in Alzheimer's disease. Nat Med. 2017 Jun;23(6):678-680. doi: 10.1038/nm.4330. Epub 2017 May 1. PMID 28459436
- [Background] Vossel KA, Beagle AJ, Rabinovici GD, Shu H, Lee SE, Naasan G, Hegde M, Cornes SB, Henry ML, Nelson AB, Seeley WW, Geschwind MD, Gorno-Tempini ML, Shih T, Kirsch HE, Garcia PA, Miller BL, Mucke L. Seizures and epileptiform activity in the early stages of Alzheimer disease. JAMA Neurol. 2013 Sep 1;70(9):1158-66. doi: 10.1001/jamaneurol.2013.136. PMID 23835471
- [Background] Vossel KA, Ranasinghe KG, Beagle AJ, Mizuiri D, Honma SM, Dowling AF, Darwish SM, Van Berlo V, Barnes DE, Mantle M, Karydas AM, Coppola G, Roberson ED, Miller BL, Garcia PA, Kirsch HE, Mucke L, Nagarajan SS. Incidence and impact of subclinical epileptiform activity in Alzheimer's disease. Ann Neurol. 2016 Dec;80(6):858-870. doi: 10.1002/ana.24794. Epub 2016 Nov 7. PMID 27696483
- [Background] Vossel KA, Tartaglia MC, Nygaard HB, Zeman AZ, Miller BL. Epileptic activity in Alzheimer's disease: causes and clinical relevance. Lancet Neurol. 2017 Apr;16(4):311-322. doi: 10.1016/S1474-4422(17)30044-3. PMID 28327340
- [Background] Lam AD, Zepeda R, Cole AJ, Cash SS. Widespread changes in network activity allow non-invasive detection of mesial temporal lobe seizures. Brain. 2016 Oct;139(Pt 10):2679-2693. doi: 10.1093/brain/aww198. Epub 2016 Jul 29. PMID 27474219
- [Background] Rabinowicz AL, Starkstein SE, Leiguarda RC, Coleman AE. Transient epileptic amnesia in dementia: a treatable unrecognized cause of episodic amnestic wandering. Alzheimer Dis Assoc Disord. 2000 Oct-Dec;14(4):231-3. doi: 10.1097/00002093-200010000-00008. PMID 11186602
- [Background] Zarea A, Charbonnier C, Rovelet-Lecrux A, Nicolas G, Rousseau S, Borden A, Pariente J, Le Ber I, Pasquier F, Formaglio M, Martinaud O, Rollin-Sillaire A, Sarazin M, Croisile B, Boutoleau-Bretonniere C, Ceccaldi M, Gabelle A, Chamard L, Blanc F, Sellal F, Paquet C, Campion D, Hannequin D, Wallon D; PHRC GMAJ Collaborators. Seizures in dominantly inherited Alzheimer disease. Neurology. 2016 Aug 30;87(9):912-9. doi: 10.1212/WNL.0000000000003048. Epub 2016 Jul 27. PMID 27466472
- [Background] Tai XY, Koepp M, Duncan JS, Fox N, Thompson P, Baxendale S, Liu JY, Reeves C, Michalak Z, Thom M. Hyperphosphorylated tau in patients with refractory epilepsy correlates with cognitive decline: a study of temporal lobe resections. Brain. 2016 Sep;139(Pt 9):2441-55. doi: 10.1093/brain/aww187. Epub 2016 Aug 7. PMID 27497924
- [Background] Horvath A, Szucs A, Barcs G, Kamondi A. Sleep EEG Detects Epileptiform Activity in Alzheimer's Disease with High Sensitivity. J Alzheimers Dis. 2017;56(3):1175-1183. doi: 10.3233/JAD-160994. PMID 28128769
- [Background] Bakker A, Krauss GL, Albert MS, Speck CL, Jones LR, Stark CE, Yassa MA, Bassett SS, Shelton AL, Gallagher M. Reduction of hippocampal hyperactivity improves cognition in amnestic mild cognitive impairment. Neuron. 2012 May 10;74(3):467-74. doi: 10.1016/j.neuron.2012.03.023. PMID 22578498
- [Background] McCurry SM, Logsdon RG, Teri L, Gibbons LE, Kukull WA, Bowen JD, McCormick WC, Larson EB. Characteristics of sleep disturbance in community-dwelling Alzheimer's disease patients. J Geriatr Psychiatry Neurol. 1999 Summer;12(2):53-9. doi: 10.1177/089198879901200203. PMID 10483925
- [Background] Ownby RL, Peruyera G, Acevedo A, Loewenstein D, Sevush S. Subtypes of sleep problems in patients with Alzheimer disease. Am J Geriatr Psychiatry. 2014 Feb;22(2):148-56. doi: 10.1016/j.jagp.2012.08.001. Epub 2013 Jan 11. PMID 23567445
- [Background] Ju YE, McLeland JS, Toedebusch CD, Xiong C, Fagan AM, Duntley SP, Morris JC, Holtzman DM. Sleep quality and preclinical Alzheimer disease. JAMA Neurol. 2013 May;70(5):587-93. doi: 10.1001/jamaneurol.2013.2334. PMID 23479184
- [Background] Pavlova M. Circadian Rhythm Sleep-Wake Disorders. Continuum (Minneap Minn). 2017 Aug;23(4, Sleep Neurology):1051-1063. doi: 10.1212/CON.0000000000000499. PMID 28777176
- [Background] Saeed Y, Abbott SM. Circadian Disruption Associated with Alzheimer's Disease. Curr Neurol Neurosci Rep. 2017 Apr;17(4):29. doi: 10.1007/s11910-017-0745-y. PMID 28324298
- [Background] Foldvary-Schaefer NR, Waters TE. Sleep-Disordered Breathing. Continuum (Minneap Minn). 2017 Aug;23(4, Sleep Neurology):1093-1116. doi: 10.1212/01.CON.0000522245.13784.f6. PMID 28777178
- [Background] Lim AS, Kowgier M, Yu L, Buchman AS, Bennett DA. Sleep Fragmentation and the Risk of Incident Alzheimer's Disease and Cognitive Decline in Older Persons. Sleep. 2013 Jul 1;36(7):1027-1032. doi: 10.5665/sleep.2802. PMID 23814339
- [Background] Lim MM, Gerstner JR, Holtzman DM. The sleep-wake cycle and Alzheimer's disease: what do we know? Neurodegener Dis Manag. 2014;4(5):351-62. doi: 10.2217/nmt.14.33. PMID 25405649
- [Background] Kang JE, Lim MM, Bateman RJ, Lee JJ, Smyth LP, Cirrito JR, Fujiki N, Nishino S, Holtzman DM. Amyloid-beta dynamics are regulated by orexin and the sleep-wake cycle. Science. 2009 Nov 13;326(5955):1005-7. doi: 10.1126/science.1180962. Epub 2009 Sep 24. PMID 19779148
- [Background] Slats D, Claassen JA, Lammers GJ, Melis RJ, Verbeek MM, Overeem S. Association between hypocretin-1 and amyloid-beta42 cerebrospinal fluid levels in Alzheimer's disease and healthy controls. Curr Alzheimer Res. 2012 Dec;9(10):1119-25. doi: 10.2174/156720512804142840. PMID 22742854
- [Background] Roh JH, Huang Y, Bero AW, Kasten T, Stewart FR, Bateman RJ, Holtzman DM. Disruption of the sleep-wake cycle and diurnal fluctuation of beta-amyloid in mice with Alzheimer's disease pathology. Sci Transl Med. 2012 Sep 5;4(150):150ra122. doi: 10.1126/scitranslmed.3004291. PMID 22956200
- [Background] Pase MP, Himali JJ, Grima NA, Beiser AS, Satizabal CL, Aparicio HJ, Thomas RJ, Gottlieb DJ, Auerbach SH, Seshadri S. Sleep architecture and the risk of incident dementia in the community. Neurology. 2017 Sep 19;89(12):1244-1250. doi: 10.1212/WNL.0000000000004373. Epub 2017 Aug 23. PMID 28835407
- [Background] Lim AS, Yu L, Kowgier M, Schneider JA, Buchman AS, Bennett DA. Modification of the relationship of the apolipoprotein E epsilon4 allele to the risk of Alzheimer disease and neurofibrillary tangle density by sleep. JAMA Neurol. 2013 Dec;70(12):1544-51. doi: 10.1001/jamaneurol.2013.4215. PMID 24145819
- [Background] Reynolds CF 3rd, Kupfer DJ, Taska LS, Hoch CC, Sewitch DE, Restifo K, Spiker DG, Zimmer B, Marin RS, Nelson J, et al. Sleep apnea in Alzheimer's dementia: correlation with mental deterioration. J Clin Psychiatry. 1985 Jul;46(7):257-61. PMID 4008448
- [Background] Ancoli-Israel S, Klauber MR, Butters N, Parker L, Kripke DF. Dementia in institutionalized elderly: relation to sleep apnea. J Am Geriatr Soc. 1991 Mar;39(3):258-63. doi: 10.1111/j.1532-5415.1991.tb01647.x. PMID 2005339
- [Background] Daulatzai MA. Evidence of neurodegeneration in obstructive sleep apnea: Relationship between obstructive sleep apnea and cognitive dysfunction in the elderly. J Neurosci Res. 2015 Dec;93(12):1778-94. doi: 10.1002/jnr.23634. Epub 2015 Aug 24. PMID 26301370
- [Background] Troussiere AC, Charley CM, Salleron J, Richard F, Delbeuck X, Derambure P, Pasquier F, Bombois S. Treatment of sleep apnoea syndrome decreases cognitive decline in patients with Alzheimer's disease. J Neurol Neurosurg Psychiatry. 2014 Dec;85(12):1405-8. doi: 10.1136/jnnp-2013-307544. Epub 2014 May 14. PMID 24828897
- [Background] Pornsriniyom D, Kim Hw, Bena J, Andrews ND, Moul D, Foldvary-Schaefer N. Effect of positive airway pressure therapy on seizure control in patients with epilepsy and obstructive sleep apnea. Epilepsy Behav. 2014 Aug;37:270-5. doi: 10.1016/j.yebeh.2014.07.005. Epub 2014 Aug 12. PMID 25117208
- [Background] Sheth SA, Aronson JP, Shafi MM, Phillips HW, Velez-Ruiz N, Walcott BP, Kwon CS, Mian MK, Dykstra AR, Cole A, Eskandar EN. Utility of foramen ovale electrodes in mesial temporal lobe epilepsy. Epilepsia. 2014 May;55(5):713-724. doi: 10.1111/epi.12571. Epub 2014 Mar 7. PMID 24605889
- [Background] Risse SC, Lampe TH, Bird TD, Nochlin D, Sumi SM, Keenan T, Cubberley L, Peskind E, Raskind MA. Myoclonus, seizures, and paratonia in Alzheimer disease. Alzheimer Dis Assoc Disord. 1990 Winter;4(4):217-25. doi: 10.1097/00002093-199040400-00003. PMID 2264979
- [Background] Ju YS, Ooms SJ, Sutphen C, Macauley SL, Zangrilli MA, Jerome G, Fagan AM, Mignot E, Zempel JM, Claassen JAHR, Holtzman DM. Slow wave sleep disruption increases cerebrospinal fluid amyloid-beta levels. Brain. 2017 Aug 1;140(8):2104-2111. doi: 10.1093/brain/awx148. PMID 28899014
- [Background] Subota A, Pham T, Jette N, Sauro K, Lorenzetti D, Holroyd-Leduc J. The association between dementia and epilepsy: A systematic review and meta-analysis. Epilepsia. 2017 Jun;58(6):962-972. doi: 10.1111/epi.13744. Epub 2017 Apr 11. PMID 28397967
- [Background] Malow A, Bowes RJ, Ross D. Relationship of temporal lobe seizures to sleep and arousal: a combined scalp-intracranial electrode study. Sleep. 2000 Mar 15;23(2):231-4. PMID 10737340
- [Background] Liedorp M, Stam CJ, van der Flier WM, Pijnenburg YA, Scheltens P. Prevalence and clinical significance of epileptiform EEG discharges in a large memory clinic cohort. Dement Geriatr Cogn Disord. 2010;29(5):432-7. doi: 10.1159/000278620. Epub 2010 May 26. PMID 20502017
- [Background] McBride AE, Shih TT, Hirsch LJ. Video-EEG monitoring in the elderly: a review of 94 patients. Epilepsia. 2002 Feb;43(2):165-9. doi: 10.1046/j.1528-1157.2002.24401.x. PMID 11903463
- [Background] Volicer L, Smith S, Volicer BJ. Effect of seizures on progression of dementia of the Alzheimer type. Dementia. 1995 Sep-Oct;6(5):258-63. doi: 10.1159/000106956. PMID 8528372
- [Background] Sanchez PE, Zhu L, Verret L, Vossel KA, Orr AG, Cirrito JR, Devidze N, Ho K, Yu GQ, Palop JJ, Mucke L. Levetiracetam suppresses neuronal network dysfunction and reverses synaptic and cognitive deficits in an Alzheimer's disease model. Proc Natl Acad Sci U S A. 2012 Oct 16;109(42):E2895-903. doi: 10.1073/pnas.1121081109. Epub 2012 Aug 6. PMID 22869752
- [Background] van Golde EG, Gutter T, de Weerd AW. Sleep disturbances in people with epilepsy; prevalence, impact and treatment. Sleep Med Rev. 2011 Dec;15(6):357-68. doi: 10.1016/j.smrv.2011.01.002. Epub 2011 Mar 24. PMID 21439869
- [Background] Manni R, Terzaghi M. Comorbidity between epilepsy and sleep disorders. Epilepsy Res. 2010 Aug;90(3):171-7. doi: 10.1016/j.eplepsyres.2010.05.006. Epub 2010 May 31. PMID 20570109
- See also: Mission Lucidity: Decoding Dementia — https://www.missionlucidity.com/